CLINICAL TRIAL: NCT02797067
Title: Rectally Administered Indomethacin to Prevent Post-ESWL-pancreatitis (RIPEP)
Brief Title: Rectal Indomethacin to Prevent Post ESWL-pancreatitis
Acronym: RIPEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ESWL-pancreatitis
Record Dates: First submitted 2016-05-29; First posted 2016-06-13 (Estimated); Results first posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-03

CONDITIONS: Pancreatitis
Keywords: Extracorporeal Shock Wave lithotripsy(ESWL); Prophylaxis; Indomethacin; Chronic pancreatitis
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indomethacin (Experimental): Subjects will be randomized to receive a 100-mg indomethacin suppository 30 min before ESWL.
  Interventions: Drug: indomethacin suppository
- Glycerin (Placebo Comparator): Subjects will be randomized to receive either a 100-mg identical-appearing placebo (glycerin suppository) 30 min before ESWL.
  Interventions: Drug: Glycerin Suppository

INTERVENTIONS:
Drug: indomethacin suppository — 100mg rectal indomethacin 30min before ESWL
  Arms: Indomethacin
Drug: Glycerin Suppository — 30min before ESWL
  Arms: Glycerin

SUMMARY:
The purpose of the study is to determine whether rectal indomethacin reduces the incidence of post-ESWL pancreatitis.

DETAILED DESCRIPTION:
It is a prospective, double-blind, randomized controlled trial. Patients with painful chronic pancreatitis and pancreatic stones (> 5 mm in diameter) who are treated with ESWL at Changhai Hospital will be randomly allocated to indomethacin or placebo therapy before the procedure.

ELIGIBILITY:
Inclusion Criteria:

* any patient with chronic pancreatitis and pancreatic stones (> 5 mm in diameter) undergoing P-ESWL
* at least 18 years old
* provides informed consent

Exclusion Criteria:

* readmitted to the hospital during the enrollment of the study
* contraindications to ESWL
* suspected or established malignancy
* pancreatic ascites
* receiving NSAIDs within 7 days
* contraindication to NSAIDs (including gastrointestinal hemorrhage within 4 weeks or renal dysfunction with serum creatinine >120 μmol/L)
* presence of coagulopathy or received anticoagulation therapy within 3 days
* acute pancreatitis within 3 days
* known active cardiovascular or cerebrovascular disease
* pregnant or breastfeeding women
* without a rectum (ie, status post-total proctocolectomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1370 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2021-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Shanghai Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qian YY, Ru N, Chen H, Zou WB, Wu H, Pan J, Li B, Xin L, Guo JY, Tang XY, Hu LH, Jin ZD, Wang D, Du YQ, Wang LW, Li ZS, Liao Z. Rectal indometacin to prevent pancreatitis after extracorporeal shock wave lithotripsy (RIPEP): a single-centre, double-blind, randomised, placebo-controlled trial. Lancet Gastroenterol Hepatol. 2022 Mar;7(3):238-244. doi: 10.1016/S2468-1253(21)00434-9. Epub 2022 Jan 25. PMID 35085482
- [Derived] Qian YY, Chen H, Tang XY, Jiang X, Qian W, Zou WB, Xin L, Li B, Qi YF, Hu LH, Zou DW, Jin ZD, Wang D, Du YQ, Wang LW, Liu F, Li ZS, Liao Z. Rectally administered indomethacin to prevent post-ESWL-pancreatitis (RIPEP): study protocol for a randomized controlled trial. Trials. 2017 Nov 2;18(1):513. doi: 10.1186/s13063-017-2250-7. PMID 29096689

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indomethacin | Glycerin
Started | 685 | 685
Completed | 685 | 685
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indomethacin | Glycerin | Total
Number analyzed (Participants) | 685 | 685 | 1370
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.85 (12.32) | 45.84 (12.43) | 45.35 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 197 | 391
  Male | 491 | 488 | 979
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 685 | 685 | 1370
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: the Incidence of Post-ESWL Pancreatitis
Description: Patients were identified as post-ESWL pancreatitis if meeting two out of three criteria: pain consistent with acute pancreatitis; amylase or lipase>3 times normal limit; characteristic findings on imaging, in according to the Revised Atlanta International consensus.
Time Frame: up to 1 months
Measure: Count of Participants; unit: Participants
Arm/Group | Indomethacin | Glycerin
Number analyzed (Participants) | 685 | 685
Participants | 60 | 84

2. Secondary Outcome: the Incidence and Severity of Asymptomatic Hyperamylasemia and Other Post-ESWL Complications
Description: Asymptomatic hyperamylasemia was defined as an increase in serum amylase compared with pre-ESWL levels and beyond the upper limit of the normal range but showing no related symptoms. Serum amylase will be measured in all study patients at 3 and 24 hours after the procedure and subsequently at clinical discretion.
  Other post-ESWL complications including bleeding, infection, steinstrasse and perforation.
  Bleeding is related to clinical evidence，the level of hemoglobin ( measured at 24 hours after the procedure and at clinical discretion) and treatments.
  Infection is related to temperature and treatment. Steinstrasse is related to abdominal pain degree and the combination of other complications.
  Perforation is related to treatment.
Time Frame: up to 1 months
Measure: Count of Participants; unit: Participants
Arm/Group | Indomethacin | Glycerin
Number analyzed (Participants) | 685 | 685
Participants
  Infection | 5 | 13
  Steinstrasse | 0 | 1
  Perforation | 0 | 1
  Asymptomatic Hyperamylasemia | 189 | 197
  Hematuria | 18 | 25
  Hematemesis | 9 | 14
  Melena | 19 | 16

3. Secondary Outcome: the Severity of Post-ESWL Pancreatitis Measured as Consensus Definitions for the Major Complications of ERCP（Endoscopic Retrograde Cholangiopancreatography ）
Description: Post-ESWL complications are also stratified as mild, moderate and severe depending mainly on the length of hospitalization and the need for invasive treatment.
Time Frame: up to 1 months
Measure: Count of Participants; unit: Participants
Arm/Group | Indomethacin | Glycerin
Number analyzed (Participants) | 685 | 685
Participants
  Mild | 59 | 79
  Moderate | 1 | 5
  Severe | 0 | 0

4. Other Pre Specified Outcome: Relative Risks in the Subgroup of Potential Risk Factors for Post -ESWL Pancreatitis Will be Assessed by SPSS（Statistical Product and Service Solutions，a Statistical Software）.
Description: Potential risk factors including sex, steatorrhea, pancreas divisum, frequent attack of acute pancreatitis (≥ 1/year), diabetes, CBD（common bile duct） stenosis, alcohol consumption, multiple stones, position (the 30°-right supine position) and shock wave frequency ≥100/min.These will be assess to determine whether the treatment effect differ in these pre-specified factors.
Time Frame: up to 1 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From administration of rectal indomethacin/glycerin suppositories to charge from hospital, up to one month
Arm/Group | Indomethacin | Glycerin
All-Cause Mortality (participants affected / at risk) | 0/685 | 0/685
Serious Adverse Events (participants affected / at risk) | 0/685 | 0/685
Other Adverse Events (participants affected / at risk) | 0/685 | 0/685

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT02797067/Prot_SAP_000.pdf